CLINICAL TRIAL: NCT04208685
Title: Evaluating Cognitive Outcomes in Down Syndrome-2
Brief Title: Evaluating Cognitive Outcomes in Down Syndrome
Acronym: ECODS-2
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0253
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As basic and behavioral science identify new ways to improve cognition and behavior in individuals with Down syndrome (DS), the lack of rigorous outcome measures represents an important problem for interpreting findings. Null findings in clinical trials could result from insensitive outcome measures, rather than ineffectiveness of treatment.

The long-term goal is to improve measurement of outcomes for children and adults with DS. Towards that goal, the investigators propose to test and refine a battery of cognitive measures that can be used in treatment studies focused on school-aged children and adults with Down syndrome. The batteries are designed to assess key domains of the DS phenotype where gaps remain in outcome measures, including attention, executive function, learning and memory, processing speed, and social cognition.

The investigators will examine the psychometric properties of measures (test-retest, validity, sensitivity to change), and to evaluate differences in the psychometric properties of measures as a function of variations in participant age, gender, degree of ID, and the participants' physical health and medical comorbidities. The investigators will evaluate at least 80 children and 50 adults with Down syndrome, per site, at five time points to evaluate key domains with a diverse and novel range of methods. This proposal aims to provide a preliminary evaluation to support the enhancement of clinical outcome measures, which ultimately will increase the accuracy in documenting improvements in the lives of children and young adults with Down syndrome.

DETAILED DESCRIPTION:
The purpose of the proposed project is to test and refine a battery of cognitive measures that can be used in treatment studies focused on Down syndrome. The battery is designed to assess several key domains of the Down syndrome cognitive phenotype where gaps remain in outcome measures, including attention, executive function, learning and memory, processing speed, and social cognition, considering comorbid conditions that can potentially interfere with the development within these cognitive domains. Although a single battery for the entire lifespan of the individual with Down syndrome has obvious appeal, the investigators have focused their effort on the school-age years so that the investigators can capture a key time point in development of these cognitive domains. Moreover, new pharmaceutical treatments are transitioning from adults to the school-age population, making the need greatest for this portion of the lifespan.

However, based on preliminary research from the ongoing study with children, a need was identified to evaluate measures with young adults with DS (ages 18-39). Supplementary funding will support the expansion of the project to include young adults with DS. Results will provide empirical guidance for refining a battery and form the foundation for a larger-scale study evaluating outcome measures.

For participants 6-17 years, at least 160 children with Down syndrome will be recruited across two sites for the study, and participants will be enrolled over four (4) years. Following pre-screening and the consent visit to determine study eligibility, children will be assessed at 6 time points. The first assessment will be the baseline testing/Time 0 visit to assess IQ. At Time 1 baseline assessments for other functioning will be completed. A two-week interval will separate Time 1 and Time 2, at which time test-retest reliability assessments will be collected. Time 3 will occur three months following Time 2 to evaluate test sensitivity to change. Time 4 will occur 3 months following Time 3 and Time 5 will occur 6 months after Time 4 to assess longitudinal changes. The time interval was selected to replicate the duration of many clinical trials.

For participants 18-35 years, at least one hundred young adults aged 18-29 years with DS will be recruited across two sites to participate in the study. Adults will participate in neuropsychology assessments at 5 time points. Parents/Caregivers will complete behavioral measures at all time points. At Time 1 baseline assessments will be completed. A two-week interval (+/- 3 days) will separate Time 1 and Time 2, when test-retest reliability assessments will be collected. Time 3 will occur three months following Time 2 (+/- 2 weeks), Time 4 will occur three months following Time 3 (+/- 2 weeks), and Time 5 will occur 6 months following Time 4 (+/- 2 weeks) to evaluate sensitivity to change, Time 6 will occur 24 months following Time 1 (+/- 4 weeks), Time 7 will occur 36 months following Time 1 (+/- 4 weeks), and Time 8 will occur 48 months following Time 1 (+/- 4 weeks) to evaluate sensitivity to change. The three and six-month time intervals were selected to replicate the duration of many clinical trials. The 12-month interval was selected to provide a time interval in which natural development should occur and allow the investigators to evaluate sensitivity to change. In this study, change will occur due to natural development, while in a clinical trial, change would be expected due to treatment. The ability to detect relatively small developmentally-based change over 12 months will allow the investigators to evaluate if the measures could detect similarly small changes in trials. Once recruitment goals are met for NIH standards for 100 young adults, aged 18-29, the study team may begin recruiting adults who are 29-35, as well.

ELIGIBILITY:
Inclusion Criteria:

* 6-35 years old at the time of consent.
* Documented diagnosis of DS.
* Nonverbal mental age of at least 36 months to complete assessment battery (per parent/caregiver/young adult self-report).
* Willingness to maintain stables dosages of current medication or ongoing treatment for the duration of the study to limit changes while evaluating outcome measures.
* Parent/caregiver/self-report that participant will be able to complete the study, including all visits.

Exclusion Criteria:

* History of blindness, deafness, or serious motor impairment

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited from clinics at Cincinnati Children's Hospital Medical Center (CCHMC), community physicians, and the Jane and Richard Thomas Center for Down Syndrome at CCHMC, as well as from the community physicians, clinics, and DS clinic at CSU. In addition, the Down Syndrome Association of Greater Cincinnati (DSAGC) and the Rocky Mountain Down Syndrome Association (RMDSA) will publicize our study through social media and their mailing lists that reaches over 12,000 families combined. Subjects may also be recruited from community programs such as baseball teams, Special Olympics, etc.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Psychometric properties of measures in the assessment battery, specifically establishing their test-retest reliability, validity, and sensitivity to change | Through study completion, an average of 4 years

SECONDARY OUTCOMES:
Psychometric properties of the measures as a function of variations in participant age, gender, and degree of ID | Through study completion, an average of 4 years
Psychometric properties of the measures as a function of variations in the participants' physical health and medical comorbidities | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Esbensen, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The shared databases and corresponding dataset generated for statistical analysis will include demographic information, standardized, experimental and computerized assessment data, and information from parent- and teacher-rating scales. The dataset will include all composite variables and scores, with no identifying information included. The data and associated documentation will be available to users only under a data sharing agreement.
  Prior to publication, findings from the project will be shared broadly at scientific meetings attended by ID researchers, especially those likely to be conducting clinical trials, such as meetings of the Down Syndrome Medical Interest Group, and International Down Syndrome Congress. In addition, the investigators will share information about the procedures freely with any investigators considering inclusion of cognitive outcome measures as a clinical endpoint.
Supporting Information: Study Protocol, SAP
Time Frame: Given the nature of data collection across multiple sites, data will only be made available upon completion of sampling and primary analyses outlined in the proposal. Data will be shared at the completion of the project according to any and all NIH guidelines. Data also will be archived in accordance with the scientific journals in which reports from the project are published.